CLINICAL TRIAL: NCT06936124
Title: A Pilot Clinical Trial Investigating Deep Brain Stimulation of the Pedunculopontine Nucleus for the Treatment of Alzheimer's Disease
Brief Title: Deep Brain Stimulation of the Pedunculopontine Nucleus for Alzheimer's Disease
Acronym: DBS-PPN-AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Alzheimer Society of Canada (Other); Brain Canada (Other)
Responsible Party: Principal Investigator, Taufik Valiante, Principal Investigator, Director of Surgical Epilepsy Program, Senior Scientist, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-5380
Record Dates: First submitted 2025-03-31; First posted 2025-04-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Deep Brain Stimulation; Pedunculopontine Nucleus; DBS-PPN; DBS
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation of the Pedunculopontine Nucleus (Experimental): The experimental intervention employs deep brain stimulation (DBS), a neuromodulation therapy involving the precise application of electrical impulses to targeted brain regions (the PPN) to modulate neural activity. The study intervention will span 12 months, with key milestones including DBS-PPN implantation, DBS activation and initial programming, and follow-up assessments at 3-month intervals. These follow-up visits will assess safety, feasibility, electrographic measures, and cognitive outcomes.
  All patient participants will receive the experimental intervention. This is the only arm in this study.
  Interventions: Procedure: Deep Brain Stimulation of the Pedunculopontine Nucleus

INTERVENTIONS:
Procedure: Deep Brain Stimulation of the Pedunculopontine Nucleus — The DBS implantation procedure targeting the PPN involves a neurosurgical operation performed under general anesthesia. During the procedure, thin electrodes are implanted in the PPN with the aid of advanced pre-operative imaging (MRI and CT scan) to confirm precise targeting. This device generates and transmits electrical impulses to the PPN, which can be adjusted to optimize therapeutic outcomes.
  Other Names: DBS; DBS-PPN

SUMMARY:
Alzheimer's disease (AD) is a brain disorder that gradually impacts cognitive functions such as memory, thinking, and daily functioning. Gamma oscillations are a type of brain activity thought to play a role in memory and cognition (thinking abilities). In AD, these oscillations are impaired - meaning they are smaller and slower than the brain waves observed in healthy individuals. Research suggests that enhancing these brain waves may help slow the progression of AD.

This research is investigating a technique called deep brain stimulation (DBS) of the pedunculopontine nucleus (PPN) as an experimental intervention. An electrode will be implanted in the PPN and deliver mild stimulation over the course of a 12-month period. As a novel intervention, the priority of the study is to determine if DBS-PPN is a safe and feasible intervention for mild-AD. Additionally, the study investigators are evaluating whether DBS-PPN can increase natural gamma oscillations in ways that improve memory and cognition. The insights from this study will guide the design of an accessible larger trial to more definitively assess how effective DBS-PPN could be as a treatment for AD.

Participants will:

* Undergo a 12-month experimental intervention involving DBS of the PPN. The procedure for implanting the DBS device takes approximately 2-3 hours under general anesthesia, followed by an overnight stay in the hospital for safety monitoring.
* Be required to attend regular appointments every 3 months from DBS implantation for the duration of the study. The follow-up visits will include safety and feasibility monitoring, brain scans (EEG and MEG), and cognitive assessments/questionnaires.
* Participants' caregiver will also complete questionnaires about their cognition, functioning, and overall health at the follow-up visits.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive neurodegenerative disorder that gradually impairs memory, cognitive abilities, and daily functioning, placing a significant burden not only on patients but also on caregivers and the healthcare system. Despite extensive research, current treatments provide only symptomatic relief without halting or reversing the disease's progression.

This study investigates a novel approach using deep brain stimulation (DBS) to target the pedunculopontine nucleus (PPN), a region involved in generating and regulating gamma oscillations across the brain. DBS is a neurosurgical procedure that utilizes stereotactic techniques to implant an electrode in a specific brain target, delivering electrical stimulation via a pulse generator. By stimulating the PPN, the study intervention aims to enhance gamma activity, potentially improving memory and cognition in AD patients. Preclinical studies have demonstrated that gamma enhancement has disease modifying effects in AD. Furthermore, DBS-PPN has shown cognitive improvements in Parkinson's dementia patients with a firmly established safety profile.

This pilot study is designed as a single-centre, single-cohort, open-label, non-randomized prospective clinical trial. The open-label nature means that both the researchers and the participants will be aware of the intervention being administered. The trial will recruit a small group of participants (N=6) with AD (amnestic subtype), to evaluate the safety, feasibility, and preliminary efficacy of DBS-PPN in treating AD. Each participant will serve as their own control, with outcome measures compared from before DBS implantation, and at regular follow-up visits over a 12-month period. The primary outcomes will focus on safety and feasibility metrics, serving to inform the design of a subsequent RCT. The secondary outcomes will assess electrophysiological (EEG and MEG) and cognitive measures, providing proof-of-concept for the potential disease-modifying effects of DBS-PPN.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 60 years old.
* Diagnosis of Alzheimer's Disease: Satisfied the diagnostic criteria of the National Institute of Aging - Alzheimer's Association criteria for probable AD.
* Clinical dementia rating scale global score of ≤ 1.
* Not taking an acetylcholinesterase inhibitor and/or memantine, or taking a stable dose for at least six months.
* Fluent in English.
* Caregiver available to participate in the study.

Exclusion Criteria:

* Pre-existing structural brain abnormalities (e.g., significant white matter disease, tumor, infarction, or intracranial hematoma).
* Other neurologic or psychiatric diagnoses, or medical comorbidities that would preclude patients from undergoing surgery.
* Non-fluent in English (it will be very difficult to conduct standard cognitive tests in English on non-fluent English speakers. In addition, language barrier is significant hurdle in providing standard care with communication and cognition being a main outcome measure).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility - Recruitment Rates | Study Initiation to End of Study Enrolment Period (36 month period)
  Determined by assessing recruitment trends. The effectiveness of recruitment strategies will be assessed by monitoring the rate at which eligible participants are enrolled.
Intervention Feasibility - Adherence to Study Protocol | Study Initiation to Final Participant Study Completion (3 years)
  To ensure procedural consistency across participants, adherence to the study protocol will be systematically monitored. Any protocol deviations will be documented and evaluated for their potential impact on study outcomes, ensuring the reliability and reproducibility of findings
Intervention Feasibility - Attrition Rates | Study Initiation to Final Participant Study Completion by (3 years)
  Participant retention will be assessed through an analysis of attrition rates, with particular attention to identifying the causes of dropout.
Intervention Feasibility - Participant Evaluation of Intervention | Participants will complete the exit interview at the final follow-up visit (month 12).
  Exit interviews will be conducted with participants and their caregivers to gather quantitative and qualitative information on their subjective experience and evaluation of the study intervention. Quantitative feedback on six items assessing satisfaction (e.g., understanding of study protocol, follow-up schedule manageability, likelihood of participating in future studies with same procedure) are measured on a a 5-point Likert scale (1 - "Very Dissatisfied" to 5 - "Very Satisfied"). Total score on quantitative items ranges from 6 - 30, with a higher score representing a more positive participant and caregiver evaluation of the study intervention.
Intervention Safety - Adverse Events (AEs) and Serious Adverse Events (SAEs) | Assessed at DBS implantation (Month 0) and at regular follow-up visits 1-month, 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  Possible adverse events (AEs), serious adverse events (SAEs), or unanticipated problems related to the DBS device, related surgery and/or stimulation will be closely monitored and managed as per standard of care and definitions and classifications set forth in the following subsections.
  An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational devices or procedures.
  An SAE is an event that:
  Led to death; Led to serious deterioration in the health of the subject Led to foetal distress, foetal death or a congenital abnormality or birth defect Could have led to death or a serious deterioration were it to recur.
Intervention Safety - AE Severity | Assessed at DBS implantation (Month 0) and at regular follow-up visits 1-month, 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  All AEs will be assessed by the study team using The Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 published by the U.S. Department of Health and Human Services (November 27, 2019) grading system. For AEs not included in the CTCAE defined grading system, the following guidelines will be used to describe severity:
  Grade 1, Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated;
  Grade 2, Moderate; minimal, local or non-invasive intervention indicated; limiting age- appropriate instrumental activities of daily life (ADL)*;
  Grade 3, Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL**;
  Grade 4, Life-threatening consequence; urgent intervention indicated; or
  Grade 5, Death related to AE.
Intervention Safety - AE Relationship to Study Intervention | Assessed at DBS implantation (Month 0) and at regular follow-up visits 1-month, 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  Team will determine AE's causality based on categories below:
  Definitely Related - There is clear evidence to suggest a causal relationship, and other possible contributing factors can be ruled out.
  Probably Related - There is evidence to suggest a causal relationship, and the influence of other factors is unlikely.
  Possibly Related - There is some evidence to suggest a causal relationship (e.g., the event occurred within a reasonable time. However, other factors may have contributed to the event (e.g., the participant's clinical condition, other concomitant events).
  Unlikely to be related - A clinical event whose temporal relationship to implantation/use of the study device makes a causal relationship improbable and in which other drugs, devices or underlying disease provides plausible explanations.
  Not Related - The AE is completely independent of implantation/use of the study device, and/or evidence exists that the event is definitely related to another etiology.
Intervention Safety - AE Outcome | Assessed at final follow-up visit 12-months post-DBS surgery, or at the last time of observation.
  The outcome of the AE will be defined according to the following:
  Recovered/ Resolved: The event has fully resolved at the end of the study*;
  Recovering/ Resolving: The event is improving but has not fully resolved at the end of the study*;
  Recovered/ Resolved with sequelae: The event has resolved, but retained pathological conditions resulting from the prior disease or injury;
  Not recovered/ not resolved: The event is ongoing at the end of the study*;
  Fatal: This event is determined to be the cause of death; and
  Unknown: Outcome information could not be obtained.

SECONDARY OUTCOMES:
Gamma Oscillation (GO) Power and Synchrony | Baseline before DBS surgery and at 1-month, 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  GO power spectral density and synchrony will be assessed using scalp EEG and MEG during DBS-PPN "on" and "off" epochs. These recordings will be collected during resting-state periods. Increases in gamma activity during the "on" state will be evaluated to determine the effectiveness of DBS-PPN in entraining GO rhythms.
Theta-Gamma Coupling During N-Back Memory Task | Baseline before DBS surgery and at 1-month, 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  Theta-gamma coupling will be measured using EEG and MEG recordings during the n-back task, which engages working memory and cognitive flexibility. Comparisons will be made between "on" and "off" states of DBS-PPN to evaluate whether stimulation enhances coupling and improves task performance. Theta-gamma coupling captures the interaction between slower theta rhythms (4-8 Hz) and faster GOs.
Working Memory Performance on N-Back Memory Task | Baseline before DBS surgery and at 1-month, 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  Working memory performance will be assessed using the n-back task during EEG and MEG recordings. Performance on the n-back task is measured by computing participants' accuracy (% of correct response) across trials, with higher measures indicating greater working memory performance.
Clinical Dementia Rating (CDR) - Sum of Boxes (CDR-SB) | Baseline before DBS surgery and at 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  Cognitive assessments will be employed to correlate the anticipated effects of DBS-PPN with improvements in cognitive performance. The CDR-SB will be used to provide a more granular assessment of cognitive and functional performance. It evaluates six domains, including memory, orientation, and problem-solving, and generates a total score that better captures subtle changes in disease severity. Each domain on the CDR is rated on a 5-point scale (0 = no impairment, 0.5 = questionable impairment, 1 = mild impairment, 2 = moderate impairment, 3 = severe impairment). The CDR-SB score is the total score across the domains and ranges from 0-18, with 18 indexing greater severity of cognitive impairment.
Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog): | Baseline before DBS surgery and at 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  The ADAS-Cog assesses task performance in cognitive domains such as memory, language, and praxis, and is sensitive to detecting cognitive changes over time. Performance on each domain is scored from 0 - 5, with 5 indexing more severe cognitive impairment. The ADAS-Cog score is a summation of scores across the domains, and ranges from 0 to 70, with higher scores indicating more severe cognitive impairment.
Montreal Cognitive Assessment (MoCA) | Baseline before DBS surgery and at 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  The MoCA is a 30-item screening tool designed to detect early cognitive impairments across multiple domains. The MoCA consists of 12 tasks, each corresponding to a specific domain of cognitive impairment. Points are allocated for correct task performance and summed to compute the MoCA score. Lower scores index more severe cognitive dysfunction. MoCA scores range from 0 to 30, and the threshold score for normal cognitive functioning is 26 or above.
Neuropsychiatric Inventory (NPI) | Baseline before DBS surgery and at 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  The NPI assesses behavioral and neuropsychiatric symptoms frequently observed in AD, such as agitation, depression, and apathy. It is administered through a structured interview with caregivers, who report on symptom presence, symptom severity (3-point scale, 1 "mild" - 3 "severe") and distress caused by symptoms (5-point scale, 0 "Not distressing at all" - 5 "Very Severely"), making it sensitive to treatment-related changes. The domain score is calculated by multiplying the distress and severity score. The total NPI score is calculated by adding all domain scores, with higher scores reflecting greater symptoms associated with AD. Total NPI score can range from 0 to 144.
Sleep Disorders Inventory (SDI) | Baseline before DBS surgery and at 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  The SDI expands upon the sleep-related item from the NPI. It captures the frequency (5-point scale, 0 "not present" - 4 "daily"), severity (4-point scale, 0 "not present" - 3 "marked), and caregiver burden of sleep disturbances through caregiver reports. The SDI Total score is calculated by multiplying the average frequency score by the average severity score. The SDI Total score ranges from 0-12, with higher scores indicating greater sleep disturbance.
Quality of Life in Alzheimer's Disease (QoL-AD) | Baseline before DBS surgery and at 3-months, 6-months, 9-months, and 12-months post-DBS surgery.
  The QoL-AD is a validated tool designed to assess quality of life in individuals with Alzheimer's disease. It consists of both patient and caregiver versions, capturing perceptions of physical health, social interaction, and emotional well-being. Each item is answered on a scale of 1 "poor" to 4 "Excellent". Scores on all 13 items are summed to compute the total QoL-AD score (ranging from 13-52), where higher scores index a greater QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Taufik A. Valiante, MD PhD FRCS, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT06936124/Prot_SAP_000.pdf